CLINICAL TRIAL: NCT00698815
Title: A Randomized Phase II Study to Assess the Efficacy of Pemetrexed or Sunitinib (NSC # 736511) or Pemetrexed Plus Sunitinib in the Second-Line Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Pemetrexed and/or Sunitinib as Second-Line Therapy in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00471; NCI-2009-00471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000589102; CALGB 30704 (Other: Alliance for Clinical Trials in Oncology); CALGB-30704 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2008-06-14; First posted 2008-06-17 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Sunitinib

ARMS (3):
- Arm I (pemetrexed) (Experimental): Patients receive pemetrexed disodium 500 mg/m^2 IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive sunitinib malate as in Arm II as third-line therapy.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium
- Arm II (sunitinib) (Experimental): Patients receive sunitinib malate at 37.5 mg PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive pemetrexed disodium as in Arm I as third-line therapy.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sunitinib Malate
- Arm III (pemetrexed and sunitinib) (Experimental): Patients receive pemetrexed disodium 500 mg/m^2 IV over 10 minutes on day 1 and sunitinib malate at 37.5 mg PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive third-line therapy at the discretion of the treating physician.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium; Drug: Sunitinib Malate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
  Arms: Arm I (pemetrexed); Arm III (pemetrexed and sunitinib)
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm II (sunitinib); Arm III (pemetrexed and sunitinib)

SUMMARY:
This randomized phase II trial studies pemetrexed disodium and sunitinib malate to compare how well they work when given alone or together as second-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether pemetrexed disodium and sunitinib malate are more effective when given alone or together in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 18 week progression-free survival rate of pemetrexed (pemetrexed disodium) alone (Arm I), sunitinib (sunitinib malate) alone (Arm II) and pemetrexed plus sunitinib (Arm III) in the second-line setting of advanced non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To compare the progression-free survival of the three arms. II. To estimate the response rate, duration of response, rate of stable disease, overall survival and to characterize the toxicity profiles of the three arms.

III. To estimate the response rate, duration of response, rate of stable disease, overall survival and toxicity of sunitinib in those patients on Arm I that receive this regimen in the third line setting.

IV. To assess vascular endothelial growth factor (VEGF) haplotypes in advanced non-small cell lung cancer.

V. To test change in tumor size at 6 weeks (after 2 cycles of therapy, typically the first evaluation point in this type of study) as an early predictor of therapeutic activity in second-line treatment of non-small cell lung cancer.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive pemetrexed disodium intravenously (IV) over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive sunitinib malate as in Arm II as third-line therapy.

ARM II: Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive pemetrexed disodium as in Arm I as third-line therapy.

ARM III: Patients receive pemetrexed disodium IV over 10 minutes on day 1 and sunitinib malate PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may then receive third-line therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 6 weeks until disease progression and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation: histologic or cytologic documentation of NSCLC
* Stage: IIIB/IV with evidence of disease progression following first-line therapy
* Tumor site: lung (non-small cell)
* No cavitary lesions
* Only one prior chemotherapy regimen in the first-line stage IIIB/IV setting is allowed; this could have been either a platinum- or non-platinum-based regimen
* First-line therapy must be completed >= 28 days before registration
* Prior adjuvant therapy is allowed provided the patient had one previous regimen in the advanced stage IIIB/IV setting
* At least 28 days from prior major surgery and at least 14 days from any prior radiotherapy before registration
* No prior inhibitors of VEGF receptor (VEGFR) (e.g., SU5416, SU6668, AZ6474, SU11248, PTK787, AZD2171, AEE-788, sorafenib); prior treatment with epidermal growth factor receptor (EGFR) inhibitors and bevacizumab is allowed, provided at least 4 weeks has elapsed
* No prior pemetrexed
* Patients must have measurable or non-measurable disease

  * Measurable disease

    * Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan
  * Non-measurable disease

    * All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly nonmeasurable lesions
  * Lesions that are considered non-measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Pregnant or nursing mothers are not eligible for this study; patients in their child bearing years must have a baseline negative pregnancy test (in the case of females); males and females must practice appropriate contraceptive measures during the period of protocol therapy and for 6 months after completion of protocol therapy; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives (Norplant), or double barrier method (diaphragm plus condom)
* No ongoing cardiac dysrhythmias, atrial fibrillation, or history of corrected QT interval (QTc interval) > 500 msec (within 2 years prior to registration); the use of agents with proarrhythmic potential (e.g., quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, flecainide) is not recommended while on protocol therapy
* Patients with class I New York Heart Association (NYHA) heart failure are eligible; patients with a history of class II NYHA heart failure are eligible, provided they meet at least one of the following criteria:

  * Patients with a history of class II heart failure who are asymptomatic on treatment
  * Patients with prior anthracycline exposure
  * Patients who have received central thoracic radiation that included the heart in the radiotherapy port
* Patients with a history of symptomatic congestive heart failure within 12 months prior to entry are not eligible
* No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft or stenting, cerebrovascular accident or transient ischemic attack within the last year
* Patients with hypertension that cannot be controlled by medications (> 150/100 mmHg despite optimal medical therapy) are not eligible
* Patients who require use of therapeutic anticoagulation for thromboembolic disease are not eligible; Note: low doses of Coumadin (up to 2 mg daily) are permitted for prophylaxis of thrombosis
* No history of venous thrombosis, pulmonary embolism, or hypercoagulopathy syndrome
* No history of pulmonary hemorrhage, bleeding diathesis, or evidence of hemoptysis; patients with blood-tinged or blood-streaked sputum will be permitted on study if the hemoptysis amounts to less than 5 mL of blood per episode and less than 10 mL of blood per 24-hour period in the best estimate of the investigator
* Patients with a history of hypothyroidism or hyperthyroidism are eligible, provided they are currently euthyroid
* None of the following within 28 days of beginning treatment: abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, serious or non-healing wound, ulcer, or bone fracture
* The use of the following specific inhibitors and inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) is not permitted; the following inhibitors of CYP3A4 are prohibited within 7 days before and during treatment with sunitinib: azole antifungals (ketoconazole, itraconazole), diltiazem, clarithromycin, erythromycin, verapamil, delavirdine, and human immunodeficiency virus (HIV) protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir); the following inducers of CYP3A4 are prohibited within 12 days before beginning and during treatment with sunitinib: rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John's Wort, efavirenz, tipranavir

  * Other inhibitors and inducers of CYP3A4 may be used if necessary, but their use is discouraged
* No symptomatic or untreated central nervous system (CNS) metastases; patients with CNS metastases must be asymptomatic, must have received definitive therapy (>= 6 weeks since resection or >= 2 weeks since radiotherapy) for brain metastases, and be off steroids or on a stable dose for 2 weeks prior to registration
* No chronic daily treatment with aspirin (> 325 mg/day) or non-steroidal antiinflammatory agents known to inhibit platelet function; treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal) is not allowed
* No pleural effusions or ascites that are detectable on physical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Heist, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (129):
- United States (129):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Arroyo Grande Community, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente Hospital, Fontana, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - PCR Oncology, Pismo Beach, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Riverside, Riverside, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente, Woodland Hills, California
  - Hartford Hospital, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Lakeland Community Hospital, Niles, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Northwell Health/Center for Advanced Medicine, New Hyde Park, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2008 and September 2011, 130 participants were recruited.
Period: Overall Study
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Started | 42 | 47 | 41
Completed | 32 | 33 | 31
Not Completed | 10 | 14 | 10
Not completed — Death | 1 | 2 | 4
Not completed — Withdrawal by Subject | 6 | 3 | 2
Not completed — MD discretion | 2 | 7 | 2
Not completed — Did not receive protocol treatment | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib) | Total
Number analyzed (Participants) | 42 | 47 | 41 | 130
Age, Customized [Number; unit: participants]
  <60 years | 16 | 15 | 15 | 46
  60-69 years | 15 | 24 | 13 | 52
  >=70 years | 11 | 8 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 19 | 61
  Male | 22 | 25 | 22 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 39 | 47 | 36 | 122
  Unknown or Not Reported | 1 | 0 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 8 | 16
  White | 36 | 43 | 32 | 111
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 47 | 41 | 130
ECOG Performance Status [Number; unit: participants] — ECOG (Eastern Cooperative Oncology Group) Performance Status is a functional impairment classification, 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2: Ambulatory and capable of all self-care but unable to carry out work activities. Up and about > 50% of waking hours; 3: Capable of limited self-care, confined to bed/chair > 50% of waking hours; 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; or 5: Dead
  participants
    0 | 13 | 17 | 14 | 44
    1 | 29 | 30 | 27 | 86
Stage (TMN) [Number; unit: participants] — The TNM staging system is based on the size and/or extent (reach) of the primary tumor (T), whether cancer cells have spread to nearby (regional) lymph nodes (N), and whether metastasis (M), or the spread of the cancer to other parts of the body, has occurred
  Stage IIIB: Extensive disease: Larger tumor size and/or spread of the cancer beyond the organ in which it first developed to nearby lymph nodes and/or tissues or organs adjacent to the location of the primary tumor Stage IV (worst): Cancer has spread to distant tissues or organs
  participants
    IIIB | 5 | 8 | 3 | 16
    IV | 37 | 39 | 38 | 114

OUTCOME MEASURES:

1. Primary Outcome: 18 Week Progression-free Survival (PFS) Rate
Description: The 18 week progression-free survival rate was defined as the proportion of patients that were alive and progression-free 18 weeks after registration into the study. Disease progression was assessed per modified RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, in either primary or nodal lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of new lesions. Kaplan-Meier estimate of 18-week progression-free survival was calculated.
Time Frame: At 18 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Number analyzed (Participants) | 42 | 47 | 41
percentage of participants | 54 [40 to 71] | 37 [25 to 54] | 48 [35 to 66]

2. Secondary Outcome: PFS
Description: PFS was defined as the time from randomization until disease progression or death, whichever occurs first. The median PFS with 95% CI was estimated using the Kaplan-Meier method. Progression is defined as in the primary outcome measure.
Time Frame: Time from randomization to disease progression and death of any cause, whichever comes first (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Number analyzed (Participants) | 42 | 47 | 41
months | 4.9 [2.1 to 8.8] | 3.3 [2.3 to 4.2] | 3.7 [2.5 to 5.8]

3. Secondary Outcome: Overall Response Rate
Description: The proportion of patients who respond (completely or partially) to each combination regimen will be estimated. An exact binomial confidence interval will be computed for these estimates.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Duration of treatment (up to 3 years)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Number analyzed (Participants) | 42 | 47 | 41
percentage of participants | 14 [5 to 29] | 17 [8 to 31] | 22 [11 to 38]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from patient randomization to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Time from randomization to death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Number analyzed (Participants) | 42 | 47 | 41
months | 10.5 [8.3 to 20.2] | 8.0 [6.8 to 13.5] | 6.7 [4.1 to 10.1]

ADVERSE EVENTS:
Description: Adverse events were evaluated for 124 participants (41, 44 and 39 on Arm I, II and III, respectively).
Arm/Group | Arm I (Pemetrexed) | Arm II (Sunitinib) | Arm III (Pemetrexed and Sunitinib)
Serious Adverse Events (participants affected / at risk) | 13/41 | 19/44 | 21/39
Other Adverse Events (participants affected / at risk) | 39/41 | 43/44 | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pemetrexed) (N=41) | Arm II (Sunitinib) (N=44) | Arm III (Pemetrexed and Sunitinib) (N=39)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (6) | 11 (13) | 13 (16)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (7) | 3 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (10) | 9 (10)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 6 (7)
Chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2)
Death NOS (General disorders) | 1 (1) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 3 (4) | 5 (5)
Fatigue (General disorders) | 8 (11) | 14 (16) | 16 (19)
Fever (General disorders) | 0 (0) | 3 (3) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (6) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 5 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (2) | 3 (3) | 10 (10)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (5) | 6 (7)
Neutrophil count decreased (Investigations) | 1 (3) | 2 (2) | 9 (10)
Platelet count decreased (Investigations) | 3 (6) | 6 (6) | 12 (14)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 5 (7) | 8 (8)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 4 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 8 (9)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 6 (9)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (2) | 6 (6) | 5 (7)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 1 (1) | 2 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3) | 2 (2)
Kidney pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pemetrexed) (N=41) | Arm II (Sunitinib) (N=44) | Arm III (Pemetrexed and Sunitinib) (N=39)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 (66) | 18 (52) | 22 (66)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (12) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (9) | 2 (3)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (4) | 0 (0)
Eye disorder (Eye disorders) | 3 (3) | 1 (1) | 1 (2)
Optic nerve edema (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (14) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 2 (13) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 3 (7) | 3 (6)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (21) | 6 (11) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 10 (25) | 16 (65) | 10 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 5 (27) | 1 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (17) | 8 (22) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 2 (9) | 2 (2) | 1 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (4) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (13) | 16 (29) | 10 (15)
Nausea (Gastrointestinal disorders) | 12 (54) | 18 (39) | 16 (35)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Proctoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (10) | 5 (12) | 6 (15)
Chest pain (General disorders) | 5 (8) | 7 (8) | 2 (2)
Chills (General disorders) | 0 (0) | 2 (8) | 1 (1)
Disease progression (General disorders) | 0 (0) | 3 (5) | 2 (3)
Edema limbs (General disorders) | 5 (15) | 3 (3) | 8 (16)
Fatigue (General disorders) | 29 (148) | 35 (119) | 29 (92)
Fever (General disorders) | 2 (3) | 1 (1) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 1 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 3 (3) | 1 (2) | 3 (4)
Pain (General disorders) | 1 (6) | 3 (3) | 2 (9)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (6)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urethral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (5) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (10) | 1 (7) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (44) | 10 (18) | 3 (7)
Alkaline phosphatase increased (Investigations) | 6 (10) | 6 (13) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 19 (54) | 12 (23) | 11 (28)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 6 (15) | 2 (2) | 3 (4)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 2 (7)
Leukocyte count decreased (Investigations) | 4 (12) | 12 (32) | 15 (45)
Lymphocyte count decreased (Investigations) | 9 (35) | 8 (23) | 10 (37)
Neutrophil count decreased (Investigations) | 9 (16) | 8 (14) | 12 (31)
Platelet count decreased (Investigations) | 4 (9) | 27 (67) | 16 (48)
Weight gain (Investigations) | 0 (0) | 1 (1) | 2 (3)
Weight loss (Investigations) | 3 (8) | 7 (10) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 9 (18) | 11 (21) | 10 (20)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (20) | 5 (8) | 9 (39)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (9) | 10 (22) | 8 (17)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (5) | 7 (10) | 3 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (19) | 8 (20) | 6 (17)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (7) | 5 (14) | 7 (10)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 4 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (23) | 14 (38) | 9 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (21) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (12) | 8 (23) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (16) | 3 (5) | 2 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (14) | 4 (19) | 1 (4)
Ataxia (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (13) | 6 (12) | 3 (5)
Dysgeusia (Nervous system disorders) | 3 (10) | 5 (29) | 5 (7)
Headache (Nervous system disorders) | 2 (3) | 6 (17) | 7 (12)
Ischemia cerebrovascular (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (4) | 1 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (5)
Neurological disorder NOS (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (13) | 1 (1) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (57) | 8 (19) | 7 (9)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (4) | 3 (3)
Confusion (Psychiatric disorders) | 1 (8) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (33) | 4 (18) | 1 (2)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (2) | 1 (2) | 2 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (9) | 5 (13) | 10 (21)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (9) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (7) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 1 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (36) | 10 (38) | 9 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (49) | 10 (27) | 9 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (7) | 3 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 2 (3) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (22) | 1 (7) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (16) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (6) | 12 (30) | 4 (9)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (11)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (20) | 8 (15) | 7 (8)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 1 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (6) | 4 (8) | 3 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (5) | 1 (1)
Flushing (Vascular disorders) | 1 (6) | 3 (22) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (34) | 10 (22) | 12 (28)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (3)
Lymphedema (Vascular disorders) | 1 (6) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less